CLINICAL TRIAL: NCT02238977
Title: Bupropion for Depression in ESRD Patients on Hemodialysis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study stopped due to difficulty recruiting
Sponsor: University of Arkansas (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 203076; R21DK097470 (NIH)
Record Dates: First submitted 2014-09-10; First posted 2014-09-12 (Estimated); Results first posted 2018-07-17 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-05

CONDITIONS: Major Depression; End Stage Renal Disease
Keywords: depression; ESRD; hemodialysis
MeSH Terms: conditions — Depressive Disorder, Major; Kidney Failure, Chronic; Depression | interventions — Fluoxetine; Bupropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluoxetine (Active Comparator): Fluoxetine up to 20 mg orally daily for 12 weeks. Flexible dosing between a minimum of 10 mg daily and 20 mg daily as tolerated.
  Interventions: Drug: Fluoxetine
- Bupropion (Experimental): Bupropion sustained release (SR) 150 mg orally twice per week
  Interventions: Drug: Bupropion

INTERVENTIONS:
Drug: Fluoxetine — Antidepressant
  Other Names: Prozac
  Arms: Fluoxetine
Drug: Bupropion — Antidepressant
  Other Names: Wellbutrin SR
  Arms: Bupropion

SUMMARY:
The proposed study will evaluate the response and remission rates for major depressive disorder (MDD) in end-stage renal disease (ESRD) patients undergoing maintenance hemodialysis (HD) treated with bupropion or fluoxetine for 12 weeks. In addition, the study will document the relative tolerability and safety, and longitudinally contrast the effects of bupropion and fluoxetine on measures of cognitive function, fatigue, inflammation, and tryptophan (TRP) and TRP catabolites in blood. It is hypothesized that both drugs will significantly reduce MDD symptoms from baseline, and be tolerable and safe, but bupropion will be associated with greater reduction in pro-inflammatory cytokines, cognitive impairment, and fatigue compared with fluoxetine.

The Specific Aims of this study are:

Aim 1: Determine the efficacy of bupropion and fluoxetine in treatment of MDD in ESRD/HD patients.

Aim 2: Determine whether longitudinal change in MDD symptoms, cognitive dysfunction, and fatigue differ between bupropion and fluoxetine.

Aim 3: Determine whether longitudinal change in MDD symptoms, cognitive dysfunction, and fatigue correlate with change in inflammation, measures of TRP availability to brain, or neurotoxic TRP metabolites.

Hypotheses:

1. Bupropion and fluoxetine will both show efficacy in treating MDD;
2. Bupropion will lead to greater improvement in cognitive dysfunction and fatigue than fluoxetine; and
3. Change in cognition and fatigue over time will correlate with change in c-reactive protein (CRP) and quinolinic acid and change in overall depression score will correlate with measures of TRP availability.

ELIGIBILITY:
Inclusion Criteria:

* age 30-70 yrs;
* have patent and non-infected arteriovenous fistula or graft;
* are receiving maintenance HD 3 times per week lasting for 3-4 hours;
* serum albumin of ≥ 3.2 g/dl, serum phosphate of <6.5 mg/dl, and serum hemoglobin of ≥9 mg/dl in consecutive two blood tests as per the National Kidney Foundation Disease Outcomes Quality Initiative (NKF KDOQI) guidelines [subjects failing screening due to blood test will be allowed to be re-screened in 30 days];
* receiving stable or maintenance dose of iron or erythropoietin-stimulating agents, statins, angiotension receptor blockers and/or angiotension converting enzyme inhibitors, phosphate binders, vitamin D receptor analogs as these agents may influence cytokines proposed in the study;
* meet the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) criteria for MDD;
* have a Ham-D score > 17

Exclusion Criteria:

* meet DSM-IV criteria for Bipolar Disorder or other psychotic disorder in the month prior to screening;
* are taking antidepressants, anti-anxiety medications, or hypnotics (including Zyban for smoking cessation);
* having failed to respond to or tolerate bupropion or fluoxetine in the past
* allergic to fluoxetine or bupropion
* known history of HIV/AIDS; No testing will be conducted for screening purposes
* known history of alcohol or drug abuse or dependence within the month prior to screening based on clinical records;
* history of myocardial infarction or heart failure within one month of screening or a history of seizures or stroke at any point;
* history of chronic liver disease and diagnosis of hepatic encephalopathy based on clinical records;
* currently diagnosed with cancer or receiving any cancer treatment;
* history of any infection within the last 2 weeks ;
* currently taking any antibiotics, anti-inflammatory, and immune-modulator agents;
* recorded noncompliance with dialysis schedules; and
* currently participating in clinical or behavioral intervention studies.
* recorded noncompliance with dialysis schedules; and
* currently participating in clinical or behavioral intervention studies

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-03-31 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fluoxetine | Bupropion
Started | 0 | 1
Completed | 0 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Due to inability to recruit subjects study was terminated. Only one subject enrolled and completed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluoxetine | Bupropion | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 | 0
  Between 18 and 65 years |  | 0 | 0
  >=65 years |  | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 0 | 0
  Male |  | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Depression Severity
Description: Depression severity as measured by the 25-item Hamilton Depression Rating Scale. The Hamilton Depression Rating Scale has proven useful for determining the level of depression before, during, and after treatment. It is based on the clinician's interview with the patient/participant and probes symptoms such as depressed mood, guilty feelings, suicide, sleep disturbances, anxiety levels and weight loss. The rater enters a number for each symptom construct that ranges from 0 (not present) to 4 (extreme symptoms). The higher the total score the more severe the depression. The scale is scored by summing the total of all items. The maximum possible total score is 66 and the minimum is 0. A score > 17 is considered compatible with a diagnosis of major depression. A score < 10 is considered clinical remission.
  The interview and scoring takes about 15 minutes.
Time Frame: up to 12 weeks
Population: Study was terminated due to inability to recruit. No subjects were recruited for Fluoxetine arm.
Measure: Number; unit: units on a scale
Arm/Group | Bupropion | Fluoxetine
Number analyzed (Participants) | 1 | 0
units on a scale | 18 |

ADVERSE EVENTS:
Time Frame: Up to 12 weeks
Description: Study was terminated due to inability to recruit. No subjects were recruited for Fluoxetine arm.
Arm/Group | Fluoxetine | Bupropion
All-Cause Mortality (participants affected / at risk) | 0/0 | 1/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-03-10): https://cdn.clinicaltrials.gov/large-docs/77/NCT02238977/Prot_SAP_000.pdf
  • Informed Consent Form (2017-03-10): https://cdn.clinicaltrials.gov/large-docs/77/NCT02238977/ICF_001.pdf